CLINICAL TRIAL: NCT01505816
Title: Visual Outcomes After Implantation of a New Refractive Toric Multifocal Intraocular Lens
Brief Title: Visual Outcomes After Implantation of a New Multifocal Intraocular Lens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, PATRICK FRENSEL DE MORAES TZELIKIS, Principal Investigator, Hospital Oftalmologico de Brasilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOB05; HOBBrasilia05 (Other: HOBBrasilia05)
Record Dates: First submitted 2012-01-03; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Cataract
Keywords: Cataract; Vision; Intraocular lens; Multifocal; Toric
MeSH Terms: conditions — Cataract | interventions — Multifocal Intraocular Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Toric (No Intervention): Multifocal Toric IOL implantation
  Interventions: Device: Multifocal Intraocular Lens (RAYNER M-FLEX T TORIC IOL)

INTERVENTIONS:
Device: Multifocal Intraocular Lens (RAYNER M-FLEX T TORIC IOL) — Multifocal IOL implantation
  Other Names: RAYNER M-FLEX T TORIC IOL

SUMMARY:
This prospective nonrandomized study comprised patients with cataract, corneal astigmatism, and motivation for spectacle independence. In all cases, a Rayner M-flex® T toric Intraocular Lens will be implanted in the capsular bag. Three months postoperatively, distance, intermediate, and near visual acuities; spherical equivalent; residual refractive astigmatism; defocus curve; and contrast sensitivity will be evaluated. A patient-satisfaction and visual phenomena questionnaire will also be administered.

DETAILED DESCRIPTION:
Postoperative evaluation was performed at 3 months. The uncorrected and corrected distance visual acuity were assessed using the 100% contrast Early Treatment Diabetic Retinopathy Study chart, uncorrected intermediate visual acuity at 70 cm, and uncorrected near visual acuity at 40 cm; a binocular defocus curve was constructed using the ETDRS chart at 4 m and adding to the patient's manifest refraction +2.50 to -5.00 D sphere in 0.50 increments. The cylinder axis of the Intraocular lens (IOL) was measured at the slitlamp using the beam protractor after full mydriasis. The mean of the absolute values of degrees the intraocular lens was off axis was determined.

Contrast sensitivity was measured using the CSV-1000 HGT instrument (VectorVision, Inc.), which presents a translucent chart divided into 4 cycles with spatial frequencies of 3, 6, 12 and 18 cycles per degree. The background illumination of the translucent chart does not depend on room lighting. All measurements were obtained under mesopic (5 cd/m2) and photopic (85 cd/m2) conditions. The examinations were performed unilaterally at a distance of 2.5 m with Best-corrected visual acuity (BCVA) and an undilated pupil. All measurements were performed under the same conditions.

Patient satisfaction and quality of life were assessed by a simple questionnaire. Patients were interviewed 3 months postoperative. Patients were asked about visual disturbances, visual lifestyle activities, spectacle use, and satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Any race
* Either gender
* Diagnosis of cataracts both eyes
* Pre-existing physical conditions that could skew visual results, such as Diabetes, Retinal detachment, Macular degeneration, or Cancer
* Subjects must have > 1.00 diopter of astigmatism

Exclusion Criteria:

* Central endothelial cell count less than 2000 cells/mm2 glaucoma or intraocular pressure greater than 21 mmHg amblyopia
* Retinal abnormalities
* Diabetes mellitus steroid or immunosuppressive treatment
* Connective tissue diseases

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Visual Performance After Implantation of a Toric Multifocal Refractive Intraocular Lens | 3 months postoperative
  Postoperative evaluation will be performed at 3 months. The uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) will be assessed using the 100% contrast ETDRS chart; a binocular defocus curve will be constructed using the ETDRS chart at 4 m.

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months
  Contrast sensitivity will be measured using the CSV-1000 HGT instrument (VectorVision, Inc.), which presents a translucent chart divided into 4 cycles with spatial frequencies of 3, 6, 12 and 18 cycles per degree (cpd). The background illumination of the translucent chart does not depend on room lighting. All measurements will be obtained under mesopic (5 cd/m2) and photopic (85 cd/m2) conditions. The examinations will be performed unilaterally at a distance of 2.5 m with BCVA and an undilated pupil. All measurements will be performed under the same conditions.
Patient satisfaction | 3 months
  Patient satisfaction and quality of life will be assessed by a simple questionnaire. Patients will be interviewed 3 months postoperative. Patients will be asked about visual disturbances, visual lifestyle activities, spectacle use, and satisfaction with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK F TZELIKIS, MD, PhD, Principal Investigator — HOSPITAL OFTALMOLOGICO BRASILIA
Locations (1):
- Hospital Oftalmologico Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Alio JL, Pinero DP, Tomas J, Plaza AB. Vector analysis of astigmatic changes after cataract surgery with implantation of a new toric multifocal intraocular lens. J Cataract Refract Surg. 2011 Jul;37(7):1217-29. doi: 10.1016/j.jcrs.2010.12.064. PMID 21700102
- [Background] Mojzis P, Pinero DP, Studeny P, Tomas J, Korda V, Plaza AB, Alio JL. Comparative analysis of clinical outcomes obtained with a new diffractive multifocal toric intraocular lens implanted through two types of corneal incision. J Refract Surg. 2011 Sep;27(9):648-57. doi: 10.3928/1081597X-20110506-01. Epub 2011 May 20. PMID 21598872
- [Result] Visser N, Nuijts RM, de Vries NE, Bauer NJ. Visual outcomes and patient satisfaction after cataract surgery with toric multifocal intraocular lens implantation. J Cataract Refract Surg. 2011 Nov;37(11):2034-42. doi: 10.1016/j.jcrs.2011.05.041. Epub 2011 Sep 22. PMID 21940140